CLINICAL TRIAL: NCT01925196
Title: Natural History and Biomarkers of C9ORF72 Amyotrophic Lateral Sclerosis and Frontotemporal Dementia
Brief Title: Natural History and Biomarkers of Amyotrophic Lateral Sclerosis and Frontotemporal Dementia Caused by the C9ORF72 Gene Mutation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130188; 13-N-0188
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-09-19

CONDITIONS: Amyotrophic Lateral Sclerosis; Frontotemporal Lobar Degeneration
Keywords: Motor Neuron Disease; Frontotemporal Dementia; Cognitive Testing; Magnetic Resonance Imaging (MRI); Transcranial Magnetic Stimulation (TMS); Natural History
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Lobar Degeneration; Motor Neuron Disease; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- C9ORF72: Participants with C9ORF72 mutation

SUMMARY:
Background:

- Some people have a mutation in the C9ORF72 gene that causes amyotrophic lateral sclerosis (ALS) or frontotemporal dementia (FTD). The mutation causes a small piece of DNA to repeat itself thousands of times. The C9ORF gene mutation mostly occurs in families. In those families, some persons have ALS and others have FTD. Occasionally the C9ORF gene mutation occurs in persons without a family history. Researchers want to understand how this gene causes different diseases. They will study how symptoms caused by the C9ORF gene develop and change over time. They will measure symptoms that occur in ALS and in FTD. In particular, they will measure strength, ability to move, thinking, and memory. They will also see if other tests are associated with progression of disease. These tests, called biomarkers, may help detect or measure C9ORF72 disease in the future.

Objectives:

- To understand how symptoms change over time in people with mutations in a gene called C9ORF72, which causes ALS and FTD.

Eligibility:

- Adults over age 18 who have this genetic mutation

Design:

* Participants will have up to 4 in-person visits and 3 telephone interviews over 3 years. Each in-person visit may take place over several days. They may be either inpatient or outpatient visits.
* At each visit, participants will undergo a series of brain, language, and behavior tests. These will include:
* Magnetic resonance imaging (MRI) of the brain. This uses magnets, radio waves, and computers to produce detailed pictures of the brain.
* Collecting spinal fluid. The clinician will make the participant s back numb and then insert a needle to collect fluid.

<TAB>- Blood samples will be taken.

<TAB>- Participants will be asked to perform several language and movement tests.

<TAB>- Small skin samples will be taken on one visit

- Between visits, participants will answer questions about their health over the phone 3 times.

DETAILED DESCRIPTION:
Objective

The primary objective of this study is to characterize the natural history of disease in patients who carry a repeat expansion in the C9ORF72 gene, which causes amyotrophic lateral sclerosis (ALS) and frontotemporal dementia (FTD). The secondary objective is to assess whether candidate biomarkers correlate with disease progression.

Study population

62 persons with a documented repeat expansion in C9ORF72 gene who have ALS, ALS-FTD, or FTD or who are carriers of the gene mutation and have a symptomatic family member.

Design

Participants will undergo a structured battery of clinical and neuropsychological tests at enrollment and at three follow-up visits to NIH to assess disease severity. During these visits, physiological, imaging, blood, and CSF for testing of candidate biomarkers will be obtained. Between visits to NIH, assessments of functional status and cognition will be carried out by phone. Participants may be seen earlier than the scheduled follow-up visit or at home if phone assessments indicate clinical deterioration.

Outcome measures

There will be three primary outcome measures, for changes in three areas of function over the first six months. The primary measure of the severity of motor clinical function will be the ALS Functional rating scale-revised (ALSFRS-R). The primary measure of the severity of cognitive function will be changes in verbal fluency score. The primary measure of the severity of behavioral dysfunction will be the caregiver assessment of the fronto-behavioral index (FBI). Secondary clinical outcomes will be the forced vital capacity (FVC) and survival. The correlation between primary and secondary clinical outcome measures and candidate biomarkers measures will be analyzed in an exploratory fashion to determine whether candidate biomarkers are predictive of disease onset or progression.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be included if they:

* Are age 18 or older
* Have a confirmed repeat expansion in the C9ORF72 gene

EXCLUSION CRITERIA:

Patients will be excluded if they

* have other major neurological or medical diseases that may cause progressive weakness or cognitive dysfunction, such as structural brain or spinal cord disease, metabolic diseases, paraneoplastic syndromes, hereditary diseases, infectious diseases, peripheral neuropathy or radiculopathy or other significant neurological abnormalities.
* require daytime ventilator support at the time of study entry
* are unable to travel to NIH at the time of study entry
* are unwilling to have follow-up visits
* are unable to understand or decline to sign the Informed Consent at the time of study entry. Participants can remain in the study (with DPA consent and participant assent) if they lose consent capacity.
* have pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye) that exclude magnetic resonance imaging
* have unstable medical conditions that, in the opinion of the investigators, prevent safe participation in this study.
* are participating in experimental treatment trials at the time of study entry or plan such participation within 6 months of entry.

Patients will not be excluded if they are receiving standard care medications for treatment of ALS and its symptoms, or are participating in non-treatment clinical research studies. Patients will be permitted to participate in experimental treatment trials after the 6 month follow-up visit.

Patients with pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye) will not be excluded but will not undergo magnetic resonance imaging or transcranial magnetic stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with C9ORF72 mutation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Verbal Fluency Score | baseline and every 6 months therafter for 3 years
  measure of the severity of cognitive function
Fronto behavioral Index (FBI) | baseline and every 6 months thereafter for 6 years
  measure of the severity of behavioral dysfunction
ALS Functional Rating Scale Revised | baseline and every 6 months therafter for 3 years
  measure of the severity of motor clinical function

CONTACTS AND LOCATIONS:
Overall Officials: Justin Y Kwan, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Krishnan G, Raitcheva D, Bartlett D, Prudencio M, McKenna-Yasek DM, Douthwright C, Oskarsson BE, Ladha S, King OD, Barmada SJ, Miller TM, Bowser R, Watts JK, Petrucelli L, Brown RH, Kankel MW, Gao FB. Poly(GR) and poly(GA) in cerebrospinal fluid as potential biomarkers for C9ORF72-ALS/FTD. Nat Commun. 2022 May 19;13(1):2799. doi: 10.1038/s41467-022-30387-4. PMID 35589711
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-N-0188.html